CLINICAL TRIAL: NCT01140438
Title: Is "Beta Cell Rest" by Insulin Treatment Beneficial Compared to State-of-the Art Enhancers of Insulin Secretion in Preserving Beta Cell Function in Subjects With Latent Autoimmune Diabetes of the Adult (LADA)?
Brief Title: Treatment of Latent Autoimmune Diabetes of the Adult
Acronym: LADA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LADA
Record Dates: First submitted 2010-06-08; First posted 2010-06-09 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Diabetes
Keywords: Latent autoimmune diabetes; adults; Beta cell rest; Insulin secretion
MeSH Terms: conditions — Diabetes Mellitus | interventions — Isophane Insulin, Human; Sitagliptin Phosphate; Metformin; repaglinide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin + NPH Insulin (Active Comparator): Patients are treated with metformin during the run-in period (3 months) and also after randomization. By randomization insulin treatment will be added in the form of injections of NPH insulin in the evenings.
  Interventions: Drug: metformin+ NPH insulin
- Metformin + sitagliptin +/-repaglinid (Active Comparator): Patients are treated with metformin during the run-in period (3 months) and also after randomization. By randomization sitagliptin tablets will be added.If HbA1c after 6 months of treatment is > 10 % above the upper limit of normal,then treatment with repaglinide tablets tree times daily at mealtimes will be added.
  Interventions: Drug: metformin + sitagliptin +/- repaglinide

INTERVENTIONS:
Drug: metformin+ NPH insulin — Metformin 500 mg + 500 mg + 1000 mg NPH insulin , initially 0.20 U/kg body weight.
  Other Names: Insulatard; Januvia
  Arms: Metformin + NPH Insulin
Drug: metformin + sitagliptin +/- repaglinide — Metformin 500 mg + 500 mg + 1000 mg Sitagliptin 100 mg x 1 Repaglinide 1 mg x 3
  Other Names: Novonorm
  Arms: Metformin + sitagliptin +/-repaglinid

SUMMARY:
The purpose of the study is to clarify whether patients classified as Latent autoimmune diabetes of the adult (LADA) benefit from early treatment with insulin added to per oral treatment and lifestyle measures.

DETAILED DESCRIPTION:
Latent autoimmune diabetes of the adult (LADA) is usually defined as a form of diabetes where the onset of diabetes takes place approximately after 30 years of age, where there is presence of beta-cell directed antibodies (mostly anti-GAD) and where there is no clinical need for insulin treatment during the first 6 months after the diagnosis of diabetes.

The aetiology and treatment of LADA patients is much less elucidated than is the case for type 1 diabetes (DM1) and type 2 diabetes (DM2). LADA constitutes about 10 % of the total diabetic population in many countries. LADA is therefore more common than insulin-requiring DM1.

LADA patients lose beta-cell function faster than patients with DM2. Residual beta-cell function in DM1 is coupled to better metabolic control with lesser degree of hyperglycemia, lesser frequency of hypoglycaemic events and lesser diabetic complications.

To retain beta-cell function in LADA patients is thus highly desirable.

There are several strategies to retain beta cell function. One therapeutic strategy is to induce some degree of "beta cell rest" by treatment with exogenous insulin. Several observations indicate that such a strategy can have beneficial effects.

This is a Scandinavian multicenter non-blinded clinical trial with 78 participants with newly diagnosed LADA. Participants will be randomized to either insulin- or per oral antidiabetic treatment. Participants will be followed up for 2 years after inclusion. Beta cell function and glycemic control will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes diagnosed during 0-3 years before entering the study.
* Age > or equal to 30 years < or equal to 75 years
* anti-GAD positivity
* fasting C-peptide > or equal to 0,3 ng/ml
* no need for insulin treatment by clinical judgement for at least 3 months following the diagnosis of diabetes.
* HbA1c > 15 % above the upper limit of normal

Exclusion Criteria:

* Renal insufficiency (plasma creatinine > 150 mol/L)
* Severe retinopathy (proliferative or pre-proliferative)
* Severe cardiac disease (NYHA III-IV)
* Chronic severe illness judged by the investigator
* Females of reproductive age who wish to become pregnant during the study

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
insulin secretion | 2 years
  insulin secretion measured by fasting and glucagon-stimulated C-peptide

SECONDARY OUTCOMES:
glycemic control | 2 years
  glycemic control (HbA1c)

CONTACTS AND LOCATIONS:
Overall Officials: Valdemar Grill, med phd, Principal Investigator — Department of Cancer Research and Molecular Medicine
Locations (1):
- Valdemar Grill, Trondheim, Norway

REFERENCES:
- [Result] Hals IK, Fiskvik Fleiner H, Reimers N, Astor MC, Filipsson K, Ma Z, Grill V, Bjorklund A. Investigating optimal beta-cell-preserving treatment in latent autoimmune diabetes in adults: Results from a 21-month randomized trial. Diabetes Obes Metab. 2019 Oct;21(10):2219-2227. doi: 10.1111/dom.13797. Epub 2019 Jun 19. PMID 31148332